CLINICAL TRIAL: NCT02425579
Title: A Phase I Trial of Inhaled Carbon Monoxide for the Treatment of Sepsis-Induced Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Safety Study of Inhaled Carbon Monoxide to Treat Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Weill Medical College of Cornell University (Other); Massachusetts General Hospital (Other); Duke University (Other)
Responsible Party: Principal Investigator, Mark A. Perrella, M.D., M.D., Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1408015437
Record Dates: First submitted 2015-03-17; First posted 2015-04-24 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Inhaled Carbon Monoxide at 100 ppm for up to 90 minutes daily for 5 days
  Interventions: Drug: Inhaled Carbon Monoxide at 100ppm (4 participants)
- Cohort 1 (placebo) (Placebo Comparator): Inhaled Medical Air for up to 90 minutes daily for 5 days
  Interventions: Drug: Placebo for Inhaled Carbon Monoxide at 100ppm (2 participants)
- Cohort 2 (Experimental): Inhaled Carbon Monoxide at 200 ppm for up to 90 minutes daily for 5 days
  Interventions: Drug: Inhaled Carbon Monoxide at 200ppm (4 participants)
- Cohort 2 (Placebo) (Placebo Comparator): Inhaled Medical Air for up to 90 minutes daily for 5 days
  Interventions: Drug: Placebo for Inhaled Carbon Monoxide at 200ppm (2 participants)

INTERVENTIONS:
Drug: Inhaled Carbon Monoxide at 100ppm (4 participants) — Inhaled Carbon Monoxide at 100ppm for up to 90 minutes daily for 5 days
  Other Names: iCO
  Arms: Cohort 1
Drug: Placebo for Inhaled Carbon Monoxide at 100ppm (2 participants) — Inhaled Medical Air for up to 90 minutes daily for 5 days
  Other Names: Inhaled Medical Air
  Arms: Cohort 1 (placebo)
Drug: Inhaled Carbon Monoxide at 200ppm (4 participants) — Inhaled Carbon Monoxide at 200ppm for 90 minutes daily for 5 days
  Other Names: iCO
  Arms: Cohort 2
Drug: Placebo for Inhaled Carbon Monoxide at 200ppm (2 participants) — Inhaled Medical Air for up to 90 minutes daily for 5 days
  Other Names: Inhaled Medical Air
  Arms: Cohort 2 (Placebo)

SUMMARY:
The purpose of this study is to assess the safety of inhaled carbon monoxide (iCO) in intubated patients with sepsis-induced ARDS.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is a syndrome of severe acute lung inflammation and hypoxemic respiratory failure with an incidence of 180,000 cases annually in the U.S.Despite decades of research and recent advances in lung protective ventilator strategies, morbidity and mortality remain unacceptably high. Furthermore, no specific effective pharmacologic therapies currently exist. The lack of specific effective therapies for sepsis-related ARDS indicates a need for new treatments that target novel pathways. Carbon monoxide (CO) represents a novel therapeutic modality in ARDS based on data obtained in experimental models of ARDS and sepsis over the past decade.

CO has been shown to be protective in experimental models of Acute Lung Injury (ALI), including hyperoxia and endotoxin exposure, bleomycin, ischemia/reperfusion, and ventilator-induced lung injury (VILI). At low doses, CO has been shown to confer tissue protective effects in these ALI models. In addition, CO has been shown to decrease inflammation, enhance phagocytosis, and improve mortality in models of sepsis including endotoxemia, hemorrhagic shock, and cecal ligation and puncture (CLP). CO has also been shown to have beneficial therapeutic effects in pre-clinical models of disease including pulmonary hypertension, vascular injury, and transplantation. Furthermore, multiple human studies have demonstrated that experimental administration of several different concentrations of CO is well tolerated and that low dose inhaled CO can be safely administered to subjects in a controlled research environment.

The purpose of this study is to assess the safety of inhaled CO therapy in mechanically ventilated patients with sepsis-induced ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sepsis are defined as those with suspected or documented infection:

   Suspected or proven infection: Sites of infection include thorax, urinary tract, abdomen, skin, sinuses, central venous catheters, and central nervous system

   All eligible patients meet the new definition of sepsis (suspected or proven infection and a SOFA ≥ 2) as PaO2/FiO2 ratio < 300 = 2 SOFA points.
2. ARDS is defined when all four of the following criteria are met:

   * A PaO2/FiO2 ratio ≤ 300 with at least 5 cm H2O positive end-expiratory airway pressure (PEEP)
   * Bilateral infiltrates consistent with pulmonary edema on frontal chest radiograph
   * A need for positive pressure ventilation by an endotracheal or tracheal tube
   * No clinical evidence of left atrial hypertension for bilateral pulmonary infiltrates.
3. ARDS onset is defined as the time the last of criteria 1-4 are met. ARDS must persist through the enrollment time window of 120 hours.
4. Infiltrates considered "consistent with pulmonary edema" include any infiltrates not fully explained by mass, atelectasis, or effusion or opacities known to be chronic (greater than 1 week). Vascular redistribution, indistinct vessels, and indistinct heart borders alone are not considered "consistent with pulmonary edema" and thus would not count as qualifying opacities for this study.

Exclusion Criteria:

1. Age less than 18 years
2. Greater than 120 hours since ARDS onset
3. Pregnant or breast-feeding
4. Prisoner
5. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)
6. No consent/inability to obtain consent
7. Physician refusal to allow enrollment in the trial
8. Moribund patient not expected to survive 24 hours
9. No arterial line/no intent to place an arterial line
10. No intent/unwillingness to follow lung protective ventilation strategy
11. Severe hypoxemia defined as oxygenation saturation (SpO2) <95 or PaO2 <80 on FiO2 ≥0.8
12. Hemoglobin < 7.5 g/dl or hemoglobin < 8 g/dl and actively bleeding
13. Subjects who are Jehovah's Witnesses or are otherwise unable or unwilling to receive blood transfusions during hospitalization
14. Acute myocardial infarction (MI) or acute coronary syndrome (ACS) within the last 90 days
15. Coronary artery bypass graft (CABG) surgery within 30 days
16. Angina pectoris or use of nitrates with activities of daily living
17. Cardiopulmonary disease classified as New York Heart Association (NYHA) class IV
18. Stroke (ischemic or hemorrhagic) within the prior 3 months
19. Diffuse alveolar hemorrhage from vasculitis
20. Use of high frequency ventilation
21. Participation in other interventional studies involving investigational agents
22. Burns > 40% total body surface area
23. Use of inhaled pulmonary vasodilator therapy (eg. NO or prostaglandins)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of administration associated adverse events. | 60 Days if remains in the ICU
  1. Acute myocardial infarction (MI) within 48 hours of study drug administration
  2. Acute cerebrovascular accident (CVA) within 48 hours of study drug administration
  3. New onset atrial or ventricular arrhythmia requiring direct current (DC) cardioversion within 48 hours of study drug administration
  4. Increased oxygenation requirements defined as: an increase in fraction of inspired oxygen (FiO2) of greater than or equal to 0.2 AND increase in PEEP greater than or equal to 5 cm of water (H2O) within 6 hours of study drug administration
  5. Increase in any protocol-specified measurement of carboxyhemoglobin (COHb) greater than or equal to 10%
  6. Increase in lactate by greater than or equal to 2 mmol/L within 6 hours of study drug administration
Incidence of serious adverse events (SAEs). | 60 Days if remains in the ICU
  An SAE is any event that is fatal or immediately life threatening, is permanently disabling, or severely incapacitating, or requires or prolongs inpatient hospitalization. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered SAEs when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
Comparison between the calculated carboxyhemoglobin (COHb) level at 90 minutes using the Coburn-Forster-Kane (CFK) equation and measured COHb level at 90 minutes | 5 days
  The Coburn-Forster-Kane (CFK) equation will be used to calculate the estimated COHb level at 90 minutes for Cohorts 1 and 2.
Mean daily Sequential Organ Failure Assessment (SOFA) score | 7 days
  Organ failure will be assessed using the SOFA score. SOFA scores will be assessed daily on days 1-5, and day 7, as the SOFA score has been shown to be a reliable prognostic indicator of outcomes in critically ill patients.
Partial pressure of arterial oxygen (PaO2)/FiO2 ratio | 5 days
  PaO2/FiO2 will be measured daily on days 1-5 if a subject remains mechanically ventilated.
Oxygenation index (OI) | 5 days
  The OI will be measured daily on days 1-5 if a subject remains mechanically ventilated.
Lung injury score (LIS) | 7 Days
  The LIS is a composite 4-point scoring system including the PaO2/FiO2, PEEP, quasi-static respiratory compliance, and the extent of infiltrates on the chest X-ray. Previous randomized clinical trials in ARDS have shown that a decreased LIS correlates with improvement in lung physiology as well as important clinical outcomes including mortality and ventilator-free days (VFDs).
Vasopressor-free days | 28 days
  Ventilator-free days will be assessed on day 28.
Ventilator-free days (VFDs) | 28 days
  Ventilator-free days to day 28 are defined as the number of days from the time of initiating unassisted breathing to day 28 after randomization, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a subject returns to assisted breathing and subsequently achieves unassisted breathing to day 28, VFDs will be counted from the end of the last period of assisted breathing to day 28.
ICU-free days | 28 days
  ICU-free days will be assessed on day 28.
Hospital-free days | 60 days
  Hospital-free days will be assessed on day 60.

OTHER OUTCOMES:
Plasma biomarkers of inflammation, lung epithelial injury,endothelial injury, markers of change in other end-organ function | 5 days
  Specific Biomarkers: Plasma biomarkers of inflammation (IL-6, IL-8, IL-10, IL-1 receptor antagonist (IL-1Ra), IL-18, IL-1β, and circulating mitochondrial DNA), lung epithelial injury (RAGE), endothelial injury (vWF, Ang-2), markers of change in other end-organ function (e.g., creatinine, liver function tests, lactate)

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Fredenburgh, MD, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Weill Cornell Medical College/NewYork-Presbyterian, New York, New York
  - Duke Univesity Hospital, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fredenburgh LE, Perrella MA, Barragan-Bradford D, Hess DR, Peters E, Welty-Wolf KE, Kraft BD, Harris RS, Maurer R, Nakahira K, Oromendia C, Davies JD, Higuera A, Schiffer KT, Englert JA, Dieffenbach PB, Berlin DA, Lagambina S, Bouthot M, Sullivan AI, Nuccio PF, Kone MT, Malik MJ, Porras MAP, Finkelsztein E, Winkler T, Hurwitz S, Serhan CN, Piantadosi CA, Baron RM, Thompson BT, Choi AM. A phase I trial of low-dose inhaled carbon monoxide in sepsis-induced ARDS. JCI Insight. 2018 Dec 6;3(23):e124039. doi: 10.1172/jci.insight.124039. PMID 30518685

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT02425579/Prot_SAP_000.pdf